CLINICAL TRIAL: NCT05142852
Title: Analgesic Effect of Extracorporeal Shock Wave Therapy in Individuals With Lateral Epicondylitis: A Randomized Controlled Trial
Brief Title: Shock Wave Therapy in Individuals With Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Salameh Aldaja (Other)
Responsible Party: Sponsor-Investigator, Salameh Aldaja, Associate Professor, Isra University, Jordan
Organization: Isra University, Jordan (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17/173
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-09

CONDITIONS: Lateral Epicondylitis
Keywords: Pain; Function
MeSH Terms: conditions — Tennis Elbow; Pain | interventions — Extracorporeal Shockwave Therapy; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extracorporeal shock wave therapy (Experimental): The participants in the experiment group received 5 consecutive sessions of ESWT for 5 minutes. Treatment parameters for the shock wave therapy group were set similar to a previous study (Devrimsel et al., 2013) 2000 shock waves with 1.6 bar intensity and 16 Hz frequency were applied for five sessions using the Swiss DolorClast Master (EMS, Nyon, Switzerland). All participants used 10-cm lateral epicondyle bandages in the treatment period, while none of them received analgesic or anti-inflammatory drugs and received exercise programs.
  Interventions: Device: Extracorporeal shock wave therapy
- Conventional physiotherapy (Active Comparator): The participants in the control group received 5 sessions of conventional physical therapy intervention for 5 minutes. The control group intervention consists of a 1-minute friction massage over the common extensor tendon of the elbow, followed by 3 minutes therapeutic ultrasound with a frequency of 1.5 Hz, and a 1-minute ice massage over the common extensor tendon of the elbow. All participants used 10-cm lateral epicondyle bandages in the treatment period, while none of them received analgesic or anti-inflammatory drugs and received exercise programs.
  Interventions: Other: Conventional physiotherapy

INTERVENTIONS:
Device: Extracorporeal shock wave therapy — The participants in the experiment group received 5 consecutive sessions of ESWT for 5 minutes. Treatment parameters for the shock wave therapy group were set similar to a previous study (Devrimsel et al., 2013) 2000 shock waves with 1.6 bar intensity and 16 Hz frequency were applied for five sessions using the Swiss DolorClast Master (EMS, Nyon, Switzerland). All participants used 10-cm lateral epicondyle bandages in the treatment period, while none of them received analgesic or anti-inflammatory drugs and received exercise programs.
  Other Names: Shock wave
  Arms: Extracorporeal shock wave therapy
Other: Conventional physiotherapy — The participants in the control group received 5 sessions of conventional physical therapy intervention for 5 minutes. The control group intervention consists of a 1-minute friction massage over the common extensor tendon of the elbow, followed by 3 minutes therapeutic ultrasound with a frequency of 1.5 Hz, and a 1-minute ice massage over the common extensor tendon of the elbow. All participants used 10-cm lateral epicondyle bandages in the treatment period, while none of them received analgesic or anti-inflammatory drugs and received exercise programs.
  Other Names: Physiotherapy
  Arms: Conventional physiotherapy

SUMMARY:
A sample of 40 patients poststroke (24 males) was randomly allocated to either ESWT experimental (n=18) or conventional physiotherapy control group (n=20). All patients received 5 sessions during the treatment program. The Visual Analog Scale (VAS) and Taiwan version Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire, and dynamometer (Maximal grip strength) for each participant were assessed before and after the treatment program.

DETAILED DESCRIPTION:
The participants in the experiment group received 5 consecutive sessions of ESWT for 5 minutes. Treatment parameters for the shock wave therapy group were set similar to a previous study (Devrimsel et al., 2013) 2000 shock waves with 1.6 bar intensity and 16 Hz frequency were applied for five sessions using the Swiss DolorClast Master (EMS, Nyon, Switzerland). The participants in the control group received 5 sessions of conventional physical therapy intervention for 5 minutes. The control group intervention consists of a 1-minute friction massage over the common extensor tendon of the elbow, followed by 3 minutes therapeutic ultrasound with a frequency of 1.5 Hz, and a 1-minute ice massage over the common extensor tendon of the elbow. All participants used 10-cm lateral epicondyle bandages in the treatment period, while none of them received analgesic or anti-inflammatory drugs and received exercise programs.

ELIGIBILITY:
Inclusion Criteria:

* An inclusion criterion was a confirmed diagnosis of lateral epicondylitis with lateral elbow pain lasting more than 6 months and less than 1 year.

Exclusion Criteria:

* Participants were excluded from this study if they had cervical radiculopathy, elbow deformity, history of diabetes mellitus, hypo- or hyperthyroidism, history of malignancy, chronic inflammatory diseases, and pregnancy. Patients who received corticosteroid injections to the lateral epicondyle within 6 weeks were also excluded.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2021-06-05 (Actual); Primary Completion 2021-08-28 (Actual); Study Completion 2021-09-04 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Change from baseline Visual Analog Scale at 5 day
  Participants were asked to rate their present pain intensity, as caused by the lateral epicondylitis, from zero to 10 using the Visual Analog Scale (VAS).

SECONDARY OUTCOMES:
Upper extremity disability and symptoms | Change from baseline Upper extremity disability and symptoms at 5 day
  Upper extremity disability and symptoms were evaluated using the Taiwan version Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire (Khoury, 2009). This 30-item questionnaire asks about the participants' ability to perform 21 various tasks, includes nine questions associated with symptoms on a 5-point scale, with the score of one representing no difficulty or no symptom and the score of five representing the inability to finish the task or severe pain.
Maximal grip strength | Change from baseline maximal grip strength at 5 day
  The maximal grip strength of the involved arm was evaluated using a grip strength dynamometer (Exacta Hydraulic Hand Dynamometer, North Coast Medical Inc, Gilroy, CA). Participants were asked to grip the dynamometer as hard as possible three times at 10-second rest intervals in the sitting position, with 90 degrees of elbow flexion, the shoulder in adduction, the wrist in slight extension, and the forearm in neutral position. The highest grip strength number was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Salameh Aldaja, PhD, Principal Investigator — Isra University, Jordan
Locations (1):
- Isra University, Amman, Jordan